CLINICAL TRIAL: NCT02731183
Title: Efficacy and Safety of Fecal Microbiota Transplantation in Treatment of Chronic Intestinal Pseudo-obstruction: a Preliminary Study
Brief Title: Efficacy and Safety of Fecal Microbiota Transplantation for Chronic Intestinal Pseudo-obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Ding Chao, MD candidate, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CIPO
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Chronic Intestinal Pseudo Obstruction
Keywords: Fecal Microbiota Transplantation; Chronic intestinal pseudo obstruction; Efficacy and safety
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FMT (Experimental): Patients included will receive standard FMT, and then will be followed up for 8 weeks.
  Interventions: Procedure: fecal microbiota transplantation

INTERVENTIONS:
Procedure: fecal microbiota transplantation — Patients received frozen FMT on 6 consecutive days through nasojejunal tubes.

SUMMARY:
Chronic intestinal pseudo obstruction(CIPO) is a serious motility disorder with life-threatening condition, and it is often related with bacterial overgrowth. Fecal microbiota transplantation (FMT) results in restoration of the normal intestinal microbial community structure. The investigators planned to observe the eﬃcacy of FMT in the treatment of a series CIPO patients. Patients received FMT on 6 consecutive days through nasojejunal tubes and followed up for 8 weeks after treatment. Rate of clinical improvement and remission, feeding tolerance of enteral nutrition, CT score of intestinal obstruction, and gastrointestinal quality-of-life index(GIQLI) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients had to have a ﬁrm diagnosis diagnostic criteria for CIPO proposed by Ministry of Health, Labour, and Welfare, including documented pathological bowel dilatation on imaging in the absence of mechanical obstruction.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the tolerance of enteral nutrition (EN) through nasojejunal tube | 8 weeks
  We defined feeding intolerance (FI) as inability to deliver the amount of nutrient as a proportion of 'energy requirements', with values of 80% chosen, or a certain amount (750ml) per 24h.
the time oral intake started | 8 weeks
  The time when oral intake (both fluids and solid food) started was noted.

SECONDARY OUTCOMES:
symptomatic relief | 8 weeks
  The occurrence and severity of each of these symptoms: pain, nausea, vomiting and bloating (each scored as 0 = absent, 1 = mild, 2 = medium, 3 = severe, or 4 = could not be worse) were recorded by nurses blinded to the intervention on a daily basis.
scoring evaluation of abdominal CT | 8 weeks
  We use a computed tomography scoring system to evaluate the severity of obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China